CLINICAL TRIAL: NCT06874803
Title: Effect of "Qi-Tonifying, Yang-Warming, and Water-Resolving" Acupuncture and Moxibustion for Motor Symptom Improvement in Early Parkinson's Disease (WARMED): A Randomized Controlled Trial
Brief Title: Acupuncture and Moxibustion for Motor Symptoms in Early Parkinson's Disease
Acronym: WARMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiani Wu (Other)
Responsible Party: Sponsor-Investigator, Jiani Wu, Associate Chief Physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLCMHPP2023003
Record Dates: First submitted 2025-02-24; First posted 2025-03-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: Acupuncture; Moxibustion; Parkinson's Disease; Motor Symptoms; Rigidity
MeSH Terms: conditions — Parkinson Disease; Muscle Rigidity | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of whether they are receiving real or sham acupuncture and moxibustion.
  The treating practitioners will follow the same protocol across both groups but will remain blinded to the randomization.
  Outcome assessors and statisticians will be blinded to the group assignments during data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture and Moxibustion Group (AM) (Experimental): Participants in this group will receive acupuncture and moxibustion therapy alongside standard Parkinson's disease (PD) medication. Acupuncture at Shuifen (CV9), bilateral Yinlingquan (SP9), bilateral Zhongliao (BL33), and bilateral Weiyang (BL39), combined with moxibustion at Shuifen (CV9) and Zhongliao (BL33). Each participant will undergo treatment three times per week for eight weeks (24 total sessions). Standard PD medication will remain unchanged throughout the study.
  Interventions: Procedure: Acupuncture and Moxibustion (AM)
- Sham Acupuncture and Moxibustion Group (Sham-AM) (Sham Comparator): Participants in this group will receive sham acupuncture and sham moxibustion alongside standard PD medication. Acupuncture at non-acuipoints of bilateral Hegu (LI4) and bilateral Zusanli (ST36), with fake moxibustion at Shuifen (CV9) and bilateral Zhongliao (BL33). Treatments will be conducted three times per week for eight weeks (24 total sessions). Standard PD medication will remain unchanged.
  Interventions: Procedure: Sham Acupuncture and Moxibustion (Sham-AM)

INTERVENTIONS:
Procedure: Acupuncture and Moxibustion (AM) — Acupuncture and moxibustion group (AM): Acupuncture at Shuifen (CV9), bilateral Yinlingquan (SP9), bilateral Zhongliao (BL33), and bilateral Weiyang (BL39), combined with moxibustion at Shuifen (CV9) and Zhongliao (BL33).
  Arms: Acupuncture and Moxibustion Group (AM)
Procedure: Sham Acupuncture and Moxibustion (Sham-AM) — Sham acupuncture and moxibustion group (sham-AM): Acupuncture at non-acuipoints of bilateral Hegu (LI4) and bilateral Zusanli (ST36), with fake moxibustion at Shuifen (CV9) and bilateral Zhongliao (BL33).
  Arms: Sham Acupuncture and Moxibustion Group (Sham-AM)

SUMMARY:
This study evaluates the clinical effect and safety of acupuncture combined with moxibustion in improving motor symptoms of early-stage Parkinson's Disease (PD) patients, by assessing the changes in UPDRS scores. It also explores objective factors affecting the acupuncture effect and investigates the functional MRI mechanisms of acupuncture in PD treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Diagnosed with Parkinson's disease (PD) according to the 2016 Chinese 2. Diagnostic Criteria for Parkinson's Disease.

3. Hoehn-Yahr stage <3 (mild to moderate PD). 4. Age between 30 and 80 years (inclusive). 5. Signed informed consent indicating voluntary participation.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded:

1. Diagnosed with Parkinson-plus syndromes or other secondary parkinsonism.
2. Prior history of deep brain stimulation (DBS) surgery.
3. Severe cerebrovascular disease, brain trauma, or history of craniotomy.
4. Severe dementia or psychiatric disorders that prevent cooperation with study procedures.
5. Severe coagulation disorders.
6. Presence of severe systemic organ dysfunction (cardiac, pulmonary, hepatic, renal, endocrine, or metabolic disorders).
7. Pregnant or breastfeeding women.
8. History of allergic reaction to acupuncture or moxibustion.
9. Prior treatment with acupuncture or moxibustion within the past three months.
10. Participation in another clinical trial within the past three months.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The score change from baseline in the MDS-UPDRS part III after 8-week treatment | evaluation time points: baseline, week 8.
  The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III assesses motor function in Parkinson's disease patients. It evaluates a range of motor symptoms, including tremor, rigidity, bradykinesia, postural instability, and gait. The scale is widely used to track disease progression and response to treatment. It consists of 26 items, scored based on the severity of each symptom.

SECONDARY OUTCOMES:
The score change from baseline in the MDS-UPDRS part III after 8-week follow-up | evaluation time points: baseline, week 16.
  The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III assesses motor function in Parkinson's disease patients. It evaluates a range of motor symptoms, including tremor, rigidity, bradykinesia, postural instability, and gait. The scale is widely used to track disease progression and response to treatment. It consists of 26 items, scored based on the severity of each symptom.
Changes in VAS scores of rigidity and bradykinesia after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The VAS range from 0-10, with higher score indicating more severe symptoms
The score change from baseline in the MDS-UPDRS part II after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The MDS-UPDRS Part II evaluates the activities of daily living (ADL) in Parkinson's disease patients. It assesses how motor and non-motor symptoms impact daily functioning, including tasks such as dressing, eating, and walking. This section helps in understanding the patient's ability to perform everyday activities. It consists of 13 items, each scored based on the level of difficulty experienced.
The change from baseline in the MDS-UPDRS total score after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) is a comprehensive tool used to assess the severity of Parkinson's disease symptoms. It is divided into four parts: motor examination (Part III), activities of daily living (Part II), non-motor experiences of daily living (Part I), and motor complications (Part IV). This scale helps in tracking disease progression, evaluating treatment efficacy, and improving clinical decision-making.
The proportion of participants with ≥30% decrease of MDS-UPDRS Part III after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III assesses motor function in Parkinson's disease patients. It evaluates a range of motor symptoms, including tremor, rigidity, bradykinesia, postural instability, and gait. The scale is widely used to track disease progression and response to treatment. It consists of 26 items, scored based on the severity of each symptom.
The change from baseline in PDQ-39 after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The PDQ-39 (Parkinson's Disease Questionnaire-39) is a patient-reported outcome measure used to assess the health-related quality of life in Parkinson's disease patients. It includes 39 items covering eight domains: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and sleep. Each item is scored based on the degree of difficulty or discomfort, and the results are summarized to provide an overall score. Higher scores indicate greater impairment in quality of life.
The change from baseline in PDSS after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The Parkinson's Disease Sleep Scale (PDSS) is a tool used to assess sleep disturbances in Parkinson's disease patients. It consists of 15 items, covering sleep quality, nighttime symptoms, and daytime sleepiness. Each item is rated on a scale from 0 to 4, with higher scores indicating more severe sleep problems. The total score helps to evaluate the overall impact of sleep disturbances on the patient's quality of life.
The change from baseline in SDS after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The Self-Rating Depression Scale (SDS) is a tool used to assess the severity of depressive symptoms. It consists of 20 items, each addressing mood, behavior, and physical symptoms related to depression. Each item is scored on a 4-point scale, ranging from "none" to "severe." Higher total scores indicate more severe depressive symptoms, helping to assess the patient's mental health status.
The change from baseline in SAS after 8-week treatment and 8-week follow-up | evaluation time points: baseline, week 8, week 16.
  The Self-Rating Anxiety Scale (SAS) is a tool used to assess the severity of anxiety symptoms. It consists of 20 items, which evaluate physical and psychological symptoms of anxiety. Each item is scored on a 4-point scale, from "none" to "severe." Higher total scores indicate greater levels of anxiety, helping to gauge the patient's emotional and mental state.
The change from baseline in functional MRI signals after 8-week treatment. | evaluation time points: baseline, week 8.
  The hospital's radiology department uses functional magnetic resonance imaging (fMRI) to measure and map brain activity by detecting changes in blood oxygen level-dependent (BOLD) signals in different brain regions.
Subgroup analysis of gender in the score change from baseline in the MDS-UPDRS part III after 8-week treatment | evaluation time points: baseline, week 8.
  Stratifying by gender into male and female subgroups, we assessed the difference in MDS-UPDRS Part III scores within each subgroup to compare the efficacy between men and women. The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III assesses motor function in Parkinson's disease patients. It evaluates a range of motor symptoms, including tremor, rigidity, bradykinesia, postural instability, and gait. The scale is widely used to track disease progression and response to treatment. It consists of 26 items, scored based on the severity of each symptom.
Subgroup analysis of age in the score change from baseline in the MDS-UPDRS part III after 8-week treatment | evaluation time points: baseline, week 8.
  Age stratification was performed by dividing participants into two subgroups: those younger than 60 years and those aged 60 and above. The difference in MDS-UPDRS Part III scores was assessed within each subgroup to compare the treatment efficacy between the two age subgroups. The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III assesses motor function in Parkinson's disease patients. It evaluates a range of motor symptoms, including tremor, rigidity, bradykinesia, postural instability, and gait. The scale is widely used to track disease progression and response to treatment. It consists of 26 items, scored based on the severity of each symptom.
Subgroup analysis of disease severity in the score change from baseline in the MDS-UPDRS part III after 8-week treatment | evaluation time points: baseline, week 8.
  Patients were stratified based on disease severity using the Hoehn and Yahr staging system into four subgroups: stage 1, 1.5, 2, and 2.5. The efficacy differences across disease stages were assessed by evaluating the change in MDS-UPDRS Part III scores within each subgroup. The difference in MDS-UPDRS Part III scores was assessed within each subgroup to compare the treatment efficacy between the two age subgroups. The MDS-UPDRS (Movement Disorder Society-Unified Parkinson's Disease Rating Scale) Part III assesses motor function in Parkinson's disease patients. It evaluates a range of motor symptoms, including tremor, rigidity, bradykinesia, postural instability, and gait. The scale is widely used to track disease progression and response to treatment. It consists of 26 items, scored based on the severity of each symptom.

OTHER OUTCOMES:
The proportion of patients in intervention-related adverse events after 8-week treatment | evaluation time points: from baseline to the end of week 8.
  Acupuncture-related adverse reactions include: severe acupuncture site pain (VAS > 7), acupuncture site pain lasting more than 30 minutes, and local subcutaneous hematoma in the stimulated area. Moxibustion-related adverse reactions include: local redness and swelling, burns, and blistering. For medicines, please refer to the drug's instructions.
The proportion of patients with adherence ≥80% | evaluation time points: from baseline to the end of week 8.
  Patient adherence is assessed using the treatment frequency count method to estimate the subjects' adherence. A good adherence criterion is defined as having received 80% or more of the scheduled treatments. Adherence is calculated by dividing the number of treatments received by the number of treatments expected, multiplied by 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospita, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including all IPD that underlie the results reported in future publications. The data will include demographic information, clinical assessments, MDS-UPDRS scores, VAS scores, PDQ-39 scores, PDSS scores, SAS/SDS scores, and fMRI imaging data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be available starting 6 months after publication of the primary results and will remain accessible for at least 5 years.
Access Criteria: by email